CLINICAL TRIAL: NCT02030795
Title: Lung Deflation With Arndt® Blocker During Video-Assisted Thoracoscopy: A Comparison of the Disconnection Technique With a Continuous Bronchial Suction
Brief Title: Techniques for Lung Deflation With Arndt® Blocker
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Anesth-Dec13
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Spontaneous Pneumothorax
Keywords: Thoracic surgery; Arndt® blocker; lung deflation; Disconnection technique; Continuous suction; Elective video-assisted thoracoscopic
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Disconnection group (Active Comparator): The single lumen tube was disconnected from the ventilator for 60 s allowing the surgical lung to collapse.
  Interventions: Other: Disconnection group
- Bronchial Suction group (Active Comparator): The suction port of the bronchial blocker, and connected to -30 cm H2O of suction.
  Interventions: Other: Bronchial Suction group

INTERVENTIONS:
Other: Disconnection group — The blocker cuff was deflated, the single lumen tube was disconnected from the ventilator for 60 s allowing the surgical lung to collapse, then the cuff was re-inflated with the same amount of air as determined previously and the ventilator was reconnected to the single lumen tube
  Arms: Disconnection group
Other: Bronchial Suction group — The barrel part of a 1-mL insulin syringe was attached to the suction port of the bronchial blocker, and connected to -30 cm H2O of suction.
  Arms: Bronchial Suction group

SUMMARY:
The use of wire-guided Arndt® endobronchial blocker does not gain widespread acceptance during video-assisted thoracoscopy (VATS) because it takes longer time to collapse the operative lung especially in patients with chronic obstructive lung disease (COPD). The use of a disconnection technique for deflation of Arndt® blocker had a comparable degree of lung collapse with the use of double-lumen tubes. However, it carries a risk of blood or infected secretions contaminating the dependent lung.

We hypothesise that the use bronchial suction of through a barrel part of a 1-mL insulin syringe attached to the suction port of the bronchial blocker would be associated with comparable time to optimum lung collapse with the disconnection technique.

After ethical approval, 58 patients with spontaneous pneumothorax scheduled for elective VATS using Arndt blocker® for lung separation will be included in this prospective, randomized, double-blind study.

Patients will be randomly assigned to deflate the blocker with either disconnecting the endotracheal tube from the ventilator for 60 s. prior to inflation of the bronchial blocker allowing both lungs to collapse, or attaching -20 cm H2O of suction to the suction port of the blocker through the barrel part of a 1-mL insulin syringe (n = 29 for each group).

DETAILED DESCRIPTION:
Most Middle Eastern and British thoracic anesthesiologists (100% and 98%, respectively) are using a double-lumen endobronchial tube (DLT) as the first-choice lung separation technique, 1-2 although the intubation with a single lumen tube (SLT) could be easier. However, the use of a bronchial blocker has a special concern as it takes longer time to collapse the operative lung,3 which precludes its widespread acceptance for video-assisted thoracoscopic (VATS) procedures because of delayed insertion of the trocars.

The wire-guided Arndt® endobronchial blocker (Cook® Critical Care, Bloomington, IN) takes longer time for lung collapse than the Univent® tube (approximately, 26 min vs. 19 min, respectively; P<0.006),3 that may be due to its narrower inner lumen (1.4 mm vs. 2.0 mm, respectively).

There are different techniques described to speed of lung collapse during the use of Arndt® endobronchial blocker. These include the disconnecting of the SLT from the ventilator and allowing both lungs to collapse before inflation of the bronchial blocker cuff, 4-5 or bronchial suction either through the fiberoptic bronchoscope after deflation of the bronchial cuff and cessation of ventilation before re-inflation of the bronchial cuff, or through a barrel part of a 3-mL syringe attached to the suction port of the bronchial blocker.3 The use of a modified disconnection technique for deflation of Arndt® endobronchial blocker had a comparable degree of lung collapse with the use of DLT during VATS procedures in patients presented with pneumothorax.5 However, compared with the bronchial suction, the disconnection technique may carry a risk of blood or infected secretions contaminating the dependent lung.6

To the best of our knowledge, the comparison of the efficacy of disconnection and bronchial suction techniques to facilitate the deflation of Arndt® blocker during thoracoscopic surgery has not yet been studied.

In all patients, standard monitors and state and response entropy (SE and RE, respectively) based-depth of anaesthesia will be applied. The radial artery will be catheterized.

Anesthetic technique is standardized in all studied patients. The experienced attending anesthesiologist (>10 yrs.), who will give the anesthetic and places the Arndt® blocker will not be blinded to group assignment and will not be involved in the collection of outcome data.

After preoxygenation, anesthesia will be induced using propofol 1.5-3 mg/kg and target-controlled infusion (TCI) of remifentanil at an effect-site concentration (Ce) of 4 ng/mL, to achieve the SE values below 50 and the difference between RE and SE below 10.

Cisatracurium (0.2 mg/kg) will be given to facilitate the tracheal intubation with a SLT, size 8.0 mm for women and 8.5 mm for men. Then a 9.0 F, 78-cm Arndt® blocker will be advanced through the blocker port of its multiport adapter and the wire loop will be coupled with a pediatric fiberoptic bronchoscope (FOB) that has been introduced through the fiberoptic port. The Arndt® blocker will be introduced to the targeted bronchus. The correct position of the Arndt® blocker wil be confirmed with a FOB.

Anesthesia will be maintained with 0.7-1.5 minimum alveolar concentration (MAC) of sevoflurane and remifentanil Ce of 2-4 ng/ml to maintain the SE values below 50, the difference between RE and SE below 10 and the mean arterial blood pressure (MA) and heart rate <20% of baseline values. Cisatracurium increments will be used to maintain surgical relaxation.

Patients' two lungs (TLV) will be mechanically ventilated with fraction of inspired oxygen (FiO2) of 0.4 in air, tidal volume (VT) of 8 mL/kg, inspiratory to expiratory (I: E) ratio of 1:2.5 and PEEP of 5 cm H2O, and respiratory rate will be adjusted to achieve a PaCO2 of 35-45 mm Hg.

After the positioning of the patient in the lateral decubitus position, the position of the blocker will be reconfirmed, the blocker cuff will be inflated with a titrated amount of air to create a seal under direct visualization of FOB and the wire loop will be removed.

All surgical procedures will be performed by the same surgeons who are blinded for the lung collapse technique and who are absent from the operating room during placement of the BB and deflation of the lung.

The VATS procedure begins with the exploration of the pleural cavity using a 30° video thoracoscopic camera through a 1.5 cm single skin incision with the use of 1-3 trocars which enabled the thoracoscopic instruments to move the lung.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical class (II-III)
* Need of one lung ventilation

Exclusion Criteria:

* New York Heart Association class> II.
* Forced vital capacity (FVC) or forced expiratory volume in 1 second (FEV1) (< 50% of the predicted values).
* Severe asthma.
* Pregnancy.
* Body mass index >35 kg/m2.
* Anticipated difficult intubation.
* Patients requiring absolute lung separation.
* Known lesions along the path of the bronchial blockers.
* Need preoperative ventilatory support.
* Post-thoracic surgery pneumothorax.
* Traumatic pneumothorax.
* Emergency surgery.
* History of lung resection.
* Calculated ipsilateral percentage pneumothorax size exceeded 20% as estimated by helical CT-derived Collins'formula

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
time needed for lung collapse | 3 min before one lung ventilation
  measured from the institution of OLV to the time of total lung collapse

SECONDARY OUTCOMES:
quality of lung collapse | every 20 min intervals after one lung ventilation initiation
  The quality of lung collapse at 20 min intervals after one lung ventilation initiation according to a four-point ordinal scale,3, 8 ranging from 1 (extremely poor) to 4 (excellent). Extremely poor (Score 1) indicated no collapse; poor (Score 2) indicated that there is a partial collapse with interference with surgical exposure; good (Score 3) indicated that there is total collapse, but the lung still had residual air; and excellent (Score 4) indicated a complete collapse with perfect surgical exposure. The feasibility of this scale was investigated during six surgical procedures not included in the study.
Overall surgeon satisfaction | 15 min after surgery
  Overall surgeon satisfaction with surgical conditions as assessed using a verbal analog scale (0 = unsatisfied to 10 = very satisfied)
Number of times that the fiberoptic bronchoscope required to assure proper position | 5 min after reinflation of the surgical lung
  The number of times that the FOB was required to assure proper position or to perform further bronchial suction
Intraoperative hypoxemia | For 2 hours during surgery
  Intraoperative hypoxemia (SaO2 < 92%)

CONTACTS AND LOCATIONS:
Locations (1):
- Dammam University, Khobar, Eastern Province, Saudi Arabia

REFERENCES:
- [Derived] El-Tahan MR. A comparison of the disconnection technique with continuous bronchial suction for lung deflation when using the Arndt endobronchial blocker during video-assisted thoracoscopy: A randomised trial. Eur J Anaesthesiol. 2015 Jun;32(6):411-7. doi: 10.1097/EJA.0000000000000194. PMID 25564782